CLINICAL TRIAL: NCT07069517
Title: Accelerated Treatment for Co-occurring Insomnia, Nightmares, and PTSD: A Randomized Controlled Trial
Brief Title: Accelerated Treatment for Co-occurring Insomnia, Nightmares, and PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: The University of Texas Health Science Center at San Antonio (Other); University of Arizona (Other); NDRI-USA, Inc. (Other)
Responsible Party: Principal Investigator, Carmen McLean, Clinical Psychologist, Palo Alto Veterans Institute for Research
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MCA0010
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Insomnia; PTSD - Post Traumatic Stress Disorder; Nightmares
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Combat Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Written exposure therapy and sleep hygiene for insomnia and nightmares (Active Comparator)
  Interventions: Behavioral: Written Exposure Therapy (WET); Behavioral: Sleep Hygiene
- Written exposure therapy and CBT for insomnia and nightmares (Experimental)
  Interventions: Behavioral: Cognitive-Behavioral Therapy for Insomnia (CBTi); Behavioral: Cognitive Behavioral Therapy for Nightmares (CBTn); Behavioral: Written Exposure Therapy (WET)

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy for Insomnia (CBTi) — CBTi focuses on stimulus control, eliminating maladaptive coping habits, reducing arousal, and challenging maladaptive thoughts about sleep in an effort to reduce time to fall asleep and time awake during the night.
  Arms: Written exposure therapy and CBT for insomnia and nightmares
Behavioral: Cognitive Behavioral Therapy for Nightmares (CBTn) — CBTn involves writing about a distressing or frequent nightmare, rewriting the narrative of the nightmare to target trauma-related themes, and reading the rescripted nightmare narrative.
  Arms: Written exposure therapy and CBT for insomnia and nightmares
Behavioral: Written Exposure Therapy (WET) — WET is a trauma-focused intervention in which individuals write about their worst traumatic experience following scripted instruction from the therapist.
Behavioral: Sleep Hygiene — Involves reviewing sleep diary data, sleep education, and reviewing and discussing sleep hygiene practices.
  Arms: Written exposure therapy and sleep hygiene for insomnia and nightmares

SUMMARY:
This study is a two-arm individually randomized group treatment clinical trial evaluating behavioral therapies for insomnia, nightmares, and PTSD. The study will compare cognitive-behavioral therapy for insomnia and nightmares to sleep hygiene (Control), both integrated with Written Exposure Therapy for PTSD and delivered in an accelerated (i.e., 5-day) group treatment format, preceded and followed by individual treatment sessions. 160 participants will be randomized into one of two study conditions.

DETAILED DESCRIPTION:
The aims of the study are:

1. Determine the efficacy of accelerated cognitive behavioral therapy for insomnia and nightmares (CBTi+n) integrated with Written Exposure Therapy (WET) for PTSD for improving insomnia symptoms among military personnel with clinically significant symptoms of insomnia, nightmares, and PTSD.
2. Determine the efficacy of accelerated CBTi+n integrated with WET for improving nightmare symptoms among military personnel with clinically significant symptoms of insomnia, nightmares, and PTSD.

Exploratory Aim: Determine the efficacy of accelerated CBTi+n integrated with WET for improving PTSD symptoms among military personnel with clinically significant symptoms of insomnia, nightmares, and PTSD.

ELIGIBILITY:
Inclusion Criteria:

1. Defense Enrollment Eligibility Reporting System (DEERS) eligible active-duty military personnel or veteran, 18-65 years old.
2. Ability to speak and read English.
3. Clinically significant PTSD symptoms (CAPS-5 > 25 with at least one Intrusion symptom and at least one Avoidance symptom).
4. Clinically significant symptoms of insomnia disorder (Structured Clinical Interview for Sleep Disturbance DSM-5 (SCISD) Insomnia Criteria are met and Insomnia Severity Index (ISI) > 11).
5. Nightmares > 1 monthly (as reported on the SCISD).
6. Willing to refrain from new behavioral health or medication treatment for issues pertaining to PTSD, sleep, and nightmares during study participation.

Exclusion Criteria:

1. Current suicide or homicide risk meriting crisis intervention.
2. Inability to comprehend the baseline screening questionnaires.
3. Unwilling to remain abstinent from alcohol during therapy sessions.
4. Serious mental health symptoms, such as mania, psychosis, alcohol or substance use disorders warranting immediate clinical attention based on interviewer assessment and clinical judgement.
5. Currently engaged in evidence-based psychotherapy for PTSD (e.g., Prolonged Exposure Therapy, Cognitive Processing Therapy, Written Exposure Therapy) or insomnia or nightmares (e.g., Cognitive Behavioral Therapy for Insomnia or Nightmares).
6. Pregnancy, as determined by self-report, because pregnancy can adversely affect sleep outside of PTSD, insomnia, and nightmares.
7. Working duty shifts ending later than 21:00 or starting before 05:30 more than 2 times per month.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-12-02 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Posttraumatic Stress Disorder Checklist (PCL-5) | Change from baseline through 3 and 6 month follow-up assessment
  Self-report measure update of the PCL designed to assess PTSD symptoms as defined by the DSM-5. Total scores range from 0-80 (higher scores indicate greater PTSD severity).
Insomnia Severity Index (ISI) | Change from baseline through 3 and 6 month follow up
  The ISI assesses perceived severity of insomnia. Total scores range from 0-28 (higher scores indicate greater insomnia severity).
Nightmare Disorders Index | Change from baseline through 3 and 6 month assessments
  The NDI is a self-report assessment of nightmare disorder.

SECONDARY OUTCOMES:
Clinician Administered PTSD Scale (CAPS-5) | Change from baseline to 1-month follow-up assessment
  The CAPS-5 is a structured clinical interview that assesses the presence and severity of PTSD symptoms. Total scores range from 0-80 (higher scores indicate greater PTSD severity).
Structured Clinical Interview for DSM-5 Sleep Disorders- Revised (SCISD-R) | Change from baseline to 1-month follow-up assessment
  The SCISD-R is a semi-structured interview designed to obtain a sleep history and screen for certain sleep disorders and diagnose others, including insomnia, hypersomnia, circadian rhythm sleep-wake disorders, sleep-disordered breathing, and parasomnias.
Generalized Anxiety Disorder Screener (GAD-7) | Change from baseline through 3 and 6 month follow-up assessment
  GAD-7 is a 7-item measure that assesses generalized anxiety symptomology. Total scores range from 0-21 (higher scores indicate greater anxiety).
Trauma-Related Nightmare Survey (TRNS) | Change from baseline through 3 and 6 month follow-up assessment
  The TRNS assesses nightmare frequency, disturbance, and characteristics
Depressive Symptoms Index-Suicidality Subscale (DSI-SS) | Change from baseline through 3 and 6 month follow up assessment
  The DSI-SS is a self-report measure of suicidal ideation, plans, perceived control over ideation, and impulses for suicide. Total scores range from 0-12 (higher scores indicate greater suicidality).
Patient Health Questionnaire-9 (PHQ-9) | Change from baseline through 3 and 6 follow-up assessment
  The PHQ-9 assess the severity of affective and somatic symptoms related to depression; items correspond to the diagnostic criteria for major depression disorder. Total scores range from 0-27 (higher scores indicate greater depressive symptom severity).
Brief Inventory of Psychosocial Functioning (B-IPF) | Change from baseline through 3 and 6 month follow up
  B-IPF is a 7-item measure of functioning in seven life domains: romantic relationship, relationship with children, family relationships, friendships and socializing, work, training and education, and activities of daily living. Total scores range from 0-42 (higher scores indicate greater functional impairment).

OTHER OUTCOMES:
Neuropsychological battery | Change from second baseline to 1-month follow-up assessment
  The Neuropsychological battery draws from the from NIH toolbox Cognitive Battery and is comprised of the following tasks: Picture Vocab, Face Name Associative Memory Exam Test, Flanker Task, Oral Symbol Digit, Picture Sequence, Pattern Comparison, Dimensional Change, and Face Name Associative Memory Exam Delay.
Split Week Self-Assessment of Sleep Survey (SASS-Y) | Change from baseline through 3 and 6 month follow up assessments
  The SASS-Y measures average bedtime, sleep time, sleep onset latency, number of awakenings, wake time after sleep onset, wake time, out of bedtime and sleep quality.
Sleep Diary and Nightmare Log | Change from second baseline through to the end of treatment
  The Sleep Diary and Nightmare Log assess daily subjective sleep patterns and to inform treatment recommendations.
History of Head Injuries | Measured during baseline
  History of Head Injuries is a 3 question screener that assesses for head injury and altered consciousness.
Health Questionnaire | Measured at baseline
  Health Questionnaire measures medical and mental health diagnoses that respondents have received, medical board and disability status, medications taken, and caffeine use
Fitbit Inspire HR data will be downloaded through the Fitabase platform | Change from second baseline through 3 and 6 month follow-up
  Fitbit Inspire HR will measure heart rate, physical activity, and nighttime wakefulness.
Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) | Change from baseline through 3 and 6 month follow up assessments
  Q-SF is a 16-item measure of life satisfaction and enjoyment in different areas of life over the past week. Total scores range from 14-70 (higher scores indicate greater enjoyment and satisfaction with life).
Credibility and Expectancy Questionnaire (CEQ) | Change from pre-workshop through 1 month follow up
  The CEQ is a 6-item measure that was designed to assess treatment expectancy and rationale credibility for use in clinical outcomes studies

CONTACTS AND LOCATIONS:
Locations (1):
- Fort Hood, Kileen, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The data used to conduct these analyses are stored in the STRONG STAR Repository. Deidentified data can be accessed by emailing repository@strongstar.org